CLINICAL TRIAL: NCT05587699
Title: A Randomized, Open-label, Multiple-dose and Parallel Study to Evaluate the Pharmacokinetics, Pharmacodynamics, and Safety of CKD-843 A in Male Subjects
Brief Title: The Parallel Study to Evaluate the Pharmacokinetics, Pharmacodynamics, and Safety of CKD-843 A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A107_02PK2216
Record Dates: First submitted 2022-10-18; First posted 2022-10-20 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group - A1(Part 1) (Experimental): CKD-843 A 45mg
  Interventions: Drug: CKD-843 A 45mg(Multiple dose)
- Group - A2(Part 2) (Experimental): CKD-843 A 45mg
  Interventions: Drug: CKD-843 A 45mg
- Group - B1(Part 1) (Experimental): CKD-843 A 55mg
  Interventions: Drug: CKD-843 A 55mg(Multiple dose)
- Group - B2(Part 2) (Experimental): CKD-843 A 55mg
  Interventions: Drug: CKD-843 A 55mg
- Group - R(Part 1) (Active Comparator): CKD-843-R
  Interventions: Drug: CKD-843-R

INTERVENTIONS:
Drug: CKD-843 A 45mg(Multiple dose) — 1 Injection/3 Month, 3 times Injections
  Arms: Group - A1(Part 1)
Drug: CKD-843 A 45mg — Single Injection
  Arms: Group - A2(Part 2)
Drug: CKD-843 A 55mg(Multiple dose) — 1 Injection/3 Month, 3 times Injections
  Arms: Group - B1(Part 1)
Drug: CKD-843 A 55mg — Single Injection
  Arms: Group - B2(Part 2)
Drug: CKD-843-R — 0.5mg/day, 9 Month
  Arms: Group - R(Part 1)

SUMMARY:
A study to evaluate the pharmacokinetics, pharmacodynamics, and safety of CKD-843 A in male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Those who aged between 19 to 50
* (Part 1) Those who are diagnosed to androgenic alopecia and meet criteria BASP grade

  * M2~M3 or C2~C3 grade with V1~V3 or F1~F3
  * M1 or C1 grade with V2~V3 or F2~F3
* (Part 1) Those who consent to the condition write below

  * Scalp tattoo & to cutting hair for hair evaluation
  * Maintaining hair style & color
* (Part 2) Those who are healthy male (Regardless of alopecia)
* Those who has body weight ≥ 55kg
* Those who has calculated body mass index(BMI) of 18.5 ≤ ~ < 27.0 kg/m2

  * Body Mass Index, kg/m2= Body weight(kg)/[Height(m)2]
* Those who consent to proper contraception and do not donate sperm until 6 months after the last administration of investigational product
* Those who understanding the detailed description of this clinical trial and voluntarily decide to participate

Exclusion Criteria:

* Those who have clinically significant disease or medical history of Hepatopathy, Renal dysfunction, Neurological disorder, Immunity disorder, Respiratory disorder, Genitourinary system disorder, Hemato-oncology disorder, Cardiovascular disorder or Psychical disorder
* (Part 1) Those who meets the conditions write below

  * alopecia areata, telogen alopecia
  * Those who has psoriasis or folliculitis or scar on hair evaluation area
  * Those who has experience of platelet-enriched plasma treatment to scarp within 24 weeks before the first administration of investigational product
  * Those who has experience of light or laser treatment to scarp within 12 weeks before the first administration of investigational product
  * Those who has experience of prophylaxis or medication of hair loss within 14 days before the first administration of investigational product
* Those who take dutasteride or finasteride within 6 month before the first administration of investigational product
* Those who has hypersensitivity to dutasteride or other 5-alpha reductase related inhibitors.

  * (Part 1) Those who has hypersensitivity to tatto ink.
* Those who have the screening(D-28~D-2) test results write below

  * AST, ALT > 1.5 times higher than upper normal level
  * Total bilirubin > 1.5 times higher than upper normal level
  * eGFR (estimated Glomerular Filtration Rate, which is calculated by MDRD) < 60 mL/min/1.73m2
  * "Positive" or "Reactive" test result of Hepatitis B & C, HIV, RPR
  * Under 5 min resting condition, systolic blood pressure >150 mmHg or <90 mmHg, diastolic blood pressure >100 mmHg or <50 mmHg
* Those who has a drug abuse history within one year or positive reaction on urine drug screening test.
* Those who receive following drugs, which may affect results of clinical trial and safety Ethical-the-counter (ETC) drugs and herbal medicines within 14 days before the first administration and Over-the-counter (OTC) drugs, health foods and vitamin preparations within 7 days before the first administration of the investigational product.
* Those who take barbiturate and related (causing induction or inhibition of metabolism) drug within 30 days before the first administration of investigational product.
* Those who exceeding smoke & alcohol consumption criteria.

  * Smoke: > 10 cigarettes/day
  * Caffeine: > 5 cups/day
  * Alcohol > 210 g/week
* Those who take grapefruit within 7 days before the first administration of investigational product.
* Those who receive investigational product by participating in other clinical trial within 180 days before the first administration of investigational product.
* Those who donate whole blood within 60 days or apheresis within 30 days before the first administration of investigational product.
* Those who receive transfusion within 30 days before the first administration of investigational product.
* Those who are deemed inappropriate to participate in clinical trial by investigators.

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-10-17 (Actual)

PRIMARY OUTCOMES:
AUC0 to Day 271 | Pre-dose(Day 1 - 0 hour), Day 1 - 4 hours, Day 2, Day 8, Day 15, Day 30, Day 46, Day 61, Day 91, Day 91 - 4 hours, Day 92, Day 98, Day 105, Day 121, Day 136, Day 151, Day 181, Day 181 4 hours, Day 182, Day 188, Day 195, Day 211, Day 226, Day 241, Day 271
  Area under the concentration-time curve from time Day 1(Pre-dose) to Day 271

CONTACTS AND LOCATIONS:
Overall Officials: Minsoo Park, M.D., Ph.D, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea